CLINICAL TRIAL: NCT03793153
Title: A Novel Technique Of Uterine Cooling During Repeated Cesarean Section For Reducing Blood Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Amro M. Hetta, Doctoral Degree (MD) Candidate, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OB1
Record Dates: First submitted 2018-12-31; First posted 2019-01-04 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Cesarean Section Complications; Intrapartum Hemorrhage; Postpartum Hemorrhage; Atony, Uterine
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard Lower Segment Cesarean Section (LSCS) will be done.
- Study (Active Comparator): Uterine Cooling Technique: Standard LSCS will be done except immediately following delivery of the fetus the uterus will be externalized in the usual fashion and the body of the uterus cephalad to the hysterotomy incision will be wrapped in sterile surgical towels saturated in sterile, iced normal saline. These towels will come from a sterile cooling pot set to 30 degrees Fahrenheit. The skin of the abdomen will be draped to prevent contact with the cold towels. Iced saline-soaked towels will be kept in place for a minimum of 5 minutes and replaced at the discretion of the attending obstetrician until the hysterotomy is closed and the uterus is replaced into the patient's abdomen.
  Interventions: Procedure: Uterine Cooling Technique

INTERVENTIONS:
Procedure: Uterine Cooling Technique — Standard LSCS will be done except immediatelyfollowing delivery of the fetus the uterus will beexternalized in the usual fashion and the body of theuterus cephalad to the hysterotomy incision will bewrapped in sterile surgical towels saturated in sterile,iced normal saline. These towels will come from asterile cooling pot set to 30 degrees Fahrenheit. Theskin of the abdomen will be draped to prevent contactwith the cold towels. Iced saline-soaked towels will bekept in place for a minimum of 5 minutes and replacedat the discretion of the attending obstetrician until thehysterotomy is closed and the uterus is replaced intothe patient's abdomen.
  Other Names: Hetta-UCT
  Arms: Study

SUMMARY:
Study aim to evaluate the efficacy and safety of a novel technique of UTERINE COOLING during repeated cesarean section (CS) in reducing blood loss, and record any adverse effects following it.

DETAILED DESCRIPTION:
Bleeding during vaginal or operative delivery is always of prime concern. Despite significant progress in obstetric care 125,000 women die from obstetric hemorrhage annually in the world.

The incidence of caesarean delivery is increasing, and the average blood loss during caesarean delivery (1000 mL) is double the amount lost during vaginal delivery (500 mL).

Caesarean section (CS) rate as high as 25-30% in many areas of the world. In Egypt the CS rate is 27.6 %, in United States of America, from 1970-2009 the CS rate rose from 4.5-32.9%, and declined to 32.8% of all deliveries at 2010. In spite of the various measures to prevent blood loss during and after caesarean section, post-partum hemorrhage (PPH) continues to be the most common complication seen in almost 20% of the cases, and causes approximately 25% of maternal deaths worldwide, leading to increased maternal morbidity and mortality. Indeed we need to reduce the bleeding during and after caesarean sections aiming for reducing the morbidity and mortality rate due to obstetric hemorrhage, which can be life threatening.

The hematocrit level falls by 10% and blood transfusion is required in 6% of women undergoing caesarean delivery versus 4% of women who have a vaginal birth. Numerous methods for performing caesarean section exist targeting a safe delivery for the infant with minimum maternal morbidity. Operative morbidity includes hemorrhage, anemia, and blood products transfusion may be required associated with many risks and complications.

Women who undergo a caesarean delivery are much more likely to be delivered by a repeat operation in subsequent pregnancies. For women undergoing subsequent cesarean, the maternal risks are even greater like massive obstetric hemorrhage, hysterectomy, admission to an intensive care unit, or maternal death. Medications, such as oxytocin, misoprostol and prostaglandin F2α, have been used to control bleeding postoperatively.

The uterus is a smooth muscle whose contraction is modulated most directly by intrinsic or extrinsic oxytocin. During pregnancy the spiral arteries within the uterus and beneath the placenta enlarge to provide adequate perfusion to the placenta. After separation of the placenta the uterine smooth muscle cells contract in a pincer-like action to pinch the spiral arteries closed. When uterine contraction is inadequate (approximately 4-6% of normal pregnancies) the spiral arteries continue to bleed. If not addressed the bleeding can be excessive, even leading to maternal death. Approximately 5-8 out of 1,000 cesarean sections require hysterectomy to control bleeding.

Release of calcium ions from sarcoplasmic reticulum stores is the immediateinitiator of contraction, and calcium's diffusion from the muscle filaments andre-uptake by the sarcoplasmic reticulum results in relaxation of contraction. Insome smooth muscles cold enhances contraction; perhaps by slowing the re-uptake of calcium.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy at term between 38±5 days and 40 weeks.
* Elective planned or emergency repeated lower segment cesarean sections(LSCS).
* Pregnant women who will accept to be in the study, and have giveninformed consent.

Exclusion Criteria:

Women who refuse to be in the study, and women who are unable to consentdue to emergent nature of the cesarean section will be excluded. Women whoare unable to understand the nature of the study due to mental illness, mentalretardation, medical condition, or other communication barrier will be excluded,or who with severe medical and surgical complications as any of the followingwill be excluded :

* Heart, liver, kidney, or brain diseases, and blood disorders.
* Abruptio placenta, and placental abnormalities or accrete syndromes.
* Polyhydraminos, macrosomia, or preeclampsia.
* History of thromboembolic disorders, or severe anemia.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Intra-operative Blood Loss (ml) | 20 minutes
  Estimating Blood Loss during LSCS immediately after delivery of the fetus and prior to delivery of the placenta till closure of uterine incision.
Post-operative Vaginal Blood Loss (ml) | 6 hours
  Estimating Vaginal Blood Loss (ml) during 6 hours post LSCS.

SECONDARY OUTCOMES:
Change in Pre- versus Post-operative Hemoglobin value. | 48 hours post operative period
  Recording change in Pre- versus Post-operative Hemoglobin (g/dl) value.
Change in Pre- versus Post-operative Hematocrit value. | 48 hours post operative period
  Recording change in Pre- versus Post-operative Hematocrit (%) value.
Use of extra Oxytocin (more than 5 i.u.). | 20 minutes
  Use of extra Oxytocin (more than 5 i.u.).
Use of Methergine. | 6 hours
  Use of Methergine.
Use of Misopristole. | 6 hours
  Use of Misopristole.
Requirement of blood products. | 6 hours
  Requirement of blood products during Intra- and 6 hours Post-LSCS.
Total blood loss greater than 1000 cc. | 7 hours
  Total blood loss (ml) greater than 1000 cc.
Use of any additional measures to control blood Loss, including any pharmacological or surgical interventions. | 7 hours
  Use of any additional measures to control blood Loss, including any pharmacological or surgical interventions.
Total time uterus wrapped during hysterotomy repair. | 30 minutes
  Total time (minutes) uterus wrapped during hysterotomy repair.
Uterine temperature after wrap removal. | Less than one minute
  Uterine temperature (Fahrenheit) after wrap removal recorded by infrared thermometer.
Patient temperature pre, intra, and postoperative. | 7 hours
  Patient temperature (Fahrenheit) pre, intra, and during first 6 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Amro M. Hetta, M. Sc., Principal Investigator — OB/GYN Departments, Al-Hussein University Hospital, Al-Azhar University; Abdallah K. Ahmed, MD, Study Director — OB/GYN Departments, Al-Hussein University Hospital, Al-Azhar University; Mofeed F. Mohamed, MD, Study Chair — OB/GYN Departments, Al-Hussein University Hospital, Al-Azhar University
Locations (1):
- OB/GYN Departments, Al-Hussein University Hospital, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: After publishing
Access Criteria: Full text

REFERENCES:
- [Background] Goswami U, Sarangi S, Gupta S, Babbar S. Comparative evaluation of two doses of tranexamic acid used prophylactically in anemic parturients for lower segment cesarean section: A double-blind randomized case control prospective trial. Saudi J Anaesth. 2013 Oct;7(4):427-31. doi: 10.4103/1658-354X.121077. PMID 24348295
- [Background] Hellgren M. Hemostasis during normal pregnancy and puerperium. Semin Thromb Hemost. 2003 Apr;29(2):125-30. doi: 10.1055/s-2003-38897. PMID 12709915
- [Background] Wang HY, Hong SK, Duan Y, Yin HM. Tranexamic acid and blood loss during and after cesarean section: a meta-analysis. J Perinatol. 2015 Oct;35(10):818-25. doi: 10.1038/jp.2015.93. Epub 2015 Jul 30. PMID 26226243
- [Background] Maged AM, Helal OM, Elsherbini MM, Eid MM, Elkomy RO, Dahab S, Elsissy MH. A randomized placebo-controlled trial of preoperative tranexamic acid among women undergoing elective cesarean delivery. Int J Gynaecol Obstet. 2015 Dec;131(3):265-8. doi: 10.1016/j.ijgo.2015.05.027. Epub 2015 Aug 15. PMID 26341174
- [Background] Ahmed MR, Sayed Ahmed WA, Madny EH, Arafa AM, Said MM. Efficacy of tranexamic acid in decreasing blood loss in elective caesarean delivery. J Matern Fetal Neonatal Med. 2015 Jun;28(9):1014-8. doi: 10.3109/14767058.2014.941283. Epub 2014 Jul 28. PMID 25068947
- [Background] Movafegh A, Eslamian L, Dorabadi A. Effect of intravenous tranexamic acid administration on blood loss during and after cesarean delivery. Int J Gynaecol Obstet. 2011 Dec;115(3):224-6. doi: 10.1016/j.ijgo.2011.07.015. Epub 2011 Aug 27. PMID 21872857
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Silver RM, Landon MB, Rouse DJ, Leveno KJ, Spong CY, Thom EA, Moawad AH, Caritis SN, Harper M, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai B, Langer O, Thorp JM, Ramin SM, Mercer BM; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Maternal morbidity associated with multiple repeat cesarean deliveries. Obstet Gynecol. 2006 Jun;107(6):1226-32. doi: 10.1097/01.AOG.0000219750.79480.84. PMID 16738145
- [Background] Marshall NE, Fu R, Guise JM. Impact of multiple cesarean deliveries on maternal morbidity: a systematic review. Am J Obstet Gynecol. 2011 Sep;205(3):262.e1-8. doi: 10.1016/j.ajog.2011.06.035. Epub 2011 Jun 15. PMID 22071057
- [Background] Cahill AG, Stamilio DM, Odibo AO, Peipert JF, Ratcliffe SJ, Stevens EJ, Sammel MD, Macones GA. Is vaginal birth after cesarean (VBAC) or elective repeat cesarean safer in women with a prior vaginal delivery? Am J Obstet Gynecol. 2006 Oct;195(4):1143-7. doi: 10.1016/j.ajog.2006.06.045. Epub 2006 Jul 17. PMID 16846571
- [Background] Gungorduk K, Yildirim G, Asicioglu O, Gungorduk OC, Sudolmus S, Ark C. Efficacy of intravenous tranexamic acid in reducing blood loss after elective cesarean section: a prospective, randomized, double-blind, placebo-controlled study. Am J Perinatol. 2011 Mar;28(3):233-40. doi: 10.1055/s-0030-1268238. Epub 2010 Oct 26. PMID 20979013
- [Background] Magann EF, Evans S, Hutchinson M, Collins R, Lanneau G, Morrison JC. Postpartum hemorrhage after cesarean delivery: an analysis of risk factors. South Med J. 2005 Jul;98(7):681-5. doi: 10.1097/01.SMJ.0000163309.53317.B8. PMID 16108235
- [Background] Tarabrin O, Kaminskiy V, Galich S, Tkachenko R, Gulyaev A, Shcherbakov S, Gavrychenko D. (2012): Efficacy of tranexamic acid in decreasing blood loss during cesarean section. Critical Care, 16(Suppl 1): P439.
- [Background] World Health Organization (2010): World health report (2010) Background Paper, No 30. Available at www.who.int/entity/healthsystems/topics/financing/healthreport/30Csectioncosts.pdf.
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Wilson EC, Mathews TJ. Births: final data for 2010. Natl Vital Stat Rep. 2012 Aug 28;61(1):1-72. PMID 24974589
- [Background] World Health Organization (2006): WHO Recommendations on the Prevention of Postpartum Hemorrhage. Available at www.pphprevention.org/files/who_summaryofOct.2006techconsult.pdf.
- [Background] Gohel M, Patel P, Gupta A, Desai P. (2007): Efficacy of tranexamic acid in decreasing blood loss during and after cesarean section: A randomized case controlled prospective study. The Journal of Obstetrics and Gynecology of India, 57(3): 227-230.
- [Background] Yehia AH, Koleib MH, Abdelazim IA, Atik A. (2014): Tranexamic acid reduces blood loss during and after cesarean section: A double blinded, randomized, controlled trial. Asian Pacific Journal of Reproduction, 3(1): 53-56.
- [Background] Mitchell JL, Stecher J, Crowson J, Rich D. (2015): Uterine Cooling During Cesarean Delivery to Reduce Blood Loss and Incidence of Postpartum Hemorrhage: A Randomized Controlled Trial [79]. Obstetrics & Gynecology.